CLINICAL TRIAL: NCT00640406
Title: A Randomized, Multi-centre, Prospective Study Comparing Best Medical Treatment Versus Best Medical Treatment Plus Renal Artery Stenting in Patients With Hemodynamically Relevant Atherosclerotic Renal Artery Stenosis
Brief Title: Comparison of Best Medical Treatment Versus Best Medical Treatment Plus Renal Artery Stenting
Acronym: RADAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C0701
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STN (Experimental): Device: Dynamic Renal Stent plus Best Medical Treatment
  Interventions: Device: Dynamic Renal Stent plus Best Medical Treatment
- BMT (Active Comparator): Drug: Best Medical Treatment
  Interventions: Drug: Best Medical Treatment

INTERVENTIONS:
Device: Dynamic Renal Stent plus Best Medical Treatment — percutaneous transluminal angioplasty of the kidney artery at index procedure followed by best medical treatment for hypertension secondary to renal artery stenosis according to local standards
  Arms: STN
Drug: Best Medical Treatment — best medical treatment for hypertension secondary to renal artery stenosis according to local standards
  Arms: BMT

SUMMARY:
The clinical investigation is a prospective, international, multi-centre, randomized (1:1) trial with follow ups at 2, 6, 12 months and 3 years.

The purpose of the study is to evaluate the clinical impact of percutaneous transluminal renal artery stenting (PTRAS) on the impaired renal function measured by the estimated Glomerular Filtration Rate (eGFR) in patients with hemodynamically significant atherosclerotic renal artery stenosis (ARAS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Informed consent signed by patient (and/or legal guardian),
* Hemodynamically relevant de novo unilateral or bilateral atherosclerotic renal artery diameter stenosis RAS (≥ 70%)
* Estimated GFR > 10 ml/min calculated using the abbreviated Modification of Diet in Renal Disease (MDRD) Study equation,
* Patients presenting mild, moderate or severe hypertension (defined according to the WHO guidelines) and/or renal dysfunction,
* Target lesion must be completely coverable by one study stent,
* Total target lesion length estimated to be less than 19 mm,
* Target lesion accessible to direct stenting or, after pre-dilation, is likely to sufficiently benefit from stenting (at the discretion of the investigator),
* Renal reference vessel diameter (RVD) of ≥ 4.0 mm and < 7.0 mm based on visual estimation,
* Willingness to comply with all the specified follow-up evaluations.

Exclusion Criteria:

* Estimated GFR ≤ 10 ml/min,
* Renal atrophy or kidney length < 7cm (referring to kidney with target lesion),
* Patient not eligible for PTRAS,
* Patient not eligible for stenting,
* Target lesion occlusion,
* Target lesion and/or target vessel proximal to the target lesion is severely calcified,
* Treatment of branch lesion required,
* Fresh thrombus or embolic lesion
* Need for embolic protection in previous or planned PTRAS,
* Clotting disorders,
* INR > 2.5 before the intervention,
* Patient presents fibromuscular dysplasia,
* Prior revascularization of target lesion,
* History of target vessel revascularization within the last six months,
* Angiographic restenosis of any segment of the target vessel that has undergone prior percutaneous intervention,
* Any thrombolytic therapy procedure within 72 hours prior to planned study procedure
* Active peptic ulcer or gastro intestinal bleeding,
* Active inflammation of the kidney interfering with diagnosis and treatment of RAS (e.g. glomerulonephritis, aortitis, vasculitis),
* Radiation damage of the kidney,
* Renal disease associated with aortic aneurysm i.e. diameter of the aorta > 40 mm,
* Chronic renal replacement therapy,
* Life expectancy < 1 year,
* Co-morbid conditions limiting participation and follow-up
* Patient currently participating in another trial possibly influencing the safety of the patient and/or the outcomes of the study,
* Pregnancy/Planned pregnancy/Childbearing potential without sufficient measures to prevent pregnancy as judged by the investigator,
* Known allergy to contrast medium that cannot be adequately controlled with pre-medication,
* Known intolerance against acetylic-salicylic acid (ASA), heparin, clopidogrel and ticlopidin, cobalt-chromium,
* Metformin intake not stopped at least 48 hours before the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Difference between treatments in change of estimated glomerular filtration rate (eGFR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, PD Dr. med, Principal Investigator — Dep. of Angiology, Herzzentrum Bad Krozingen, Südring 15, 79189 Bad Krozingen, Germany
Locations (1):
- Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Zeller T, Krankenberg H, Erglis A, Blessing E, Fuss T, Scheinert D, Weser R, Doerr BB, Yollo WD, Radermacher J; RADAR Investigators. A randomized, multi-center, prospective study comparing best medical treatment versus best medical treatment plus renal artery stenting in patients with hemodynamically relevant atherosclerotic renal artery stenosis (RADAR) - one-year results of a pre-maturely terminated study. Trials. 2017 Aug 14;18(1):380. doi: 10.1186/s13063-017-2126-x. PMID 28807045
- [Derived] Schwarzwalder U, Hauk M, Zeller T. RADAR - A randomised, multi-centre, prospective study comparing best medical treatment versus best medical treatment plus renal artery stenting in patients with haemodynamically relevant atherosclerotic renal artery stenosis. Trials. 2009 Jul 27;10:60. doi: 10.1186/1745-6215-10-60. PMID 19635148